CLINICAL TRIAL: NCT00962715
Title: A Randomized, Phase I/II Clinical Trial Evaluating the Safety, Reactogenicity, and Immunogenicity of Licensed Trivalent Influenza Vaccine Administered With Recombinant Interferon Alpha Among Patients With Chronic Lymphocytic Leukemia
Brief Title: Reactogenicity, Immunogenicity of Trivalent Influenza Vaccine With Recombinant Interferon Alpha Among Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0145
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Leukemia; CLL; Influenza Vaccine Trivalent Inactivated; TIV; Flu; Pegasys; Pegylated interferon; Roferon; Interferon
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Influenza, Human | interventions — peginterferon alfa-2a; Interferons; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TIV (Experimental): TIV (Influenza Vaccine Trivalent Inactivated) alone
  Interventions: Biological: Influenza Vaccine Trivalent Inactivated (TIV)
- TIV + PEGrIFN-α (Experimental): TIV + Pegylated Interferon
  Interventions: Biological: Influenza Vaccine Trivalent Inactivated (TIV); Drug: Pegylated interferon (PEGrIFN-α, Pegasys)
- TIV + IFNα (Experimental): TIV + Interferon
  Interventions: Biological: Influenza Vaccine Trivalent Inactivated (TIV); Drug: Interferon (IFNα, Roferon-A)

INTERVENTIONS:
Biological: Influenza Vaccine Trivalent Inactivated (TIV) — 15 μg (0.5 ml) through needle into arm muscle on Days 1 and 28.
Drug: Pegylated interferon (PEGrIFN-α, Pegasys) — 180 μg (0.5 ml) before receiving TIV, through a needle under the skin.
  Other Names: Pegasys; Peginterferon alfa-2a
  Arms: TIV + PEGrIFN-α
Drug: Interferon (IFNα, Roferon-A) — 3 million units (0.5 ml) before receiving TIV, through a needle under the skin.
  Other Names: Roferon-A; Interferon alfa-2a
  Arms: TIV + IFNα

SUMMARY:
The goal of this clinical study is to learn if Pegasys (pegylated interferon) or Roferon (interferon) can make the Trivalent Inactivated Influenza vaccine (TIV) more effective in increasing the body's immune reaction against the flu virus in patients with Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
The Study Drugs:

Pegylated interferon and interferon are designed to stop the growth of viruses. Pegylated interferon has a molecule that makes it last longer in the body. Standard interferon does not have this molecule that makes it last longer.

TIV is designed to prevent the flu.

Screening Test:

Before you can start treatment on this study, you will have a "screening test" to help the doctor decide if you are eligible to take part in this study. Blood (about 4 teaspoons) will be drawn for routine tests. If you have had a routine blood test in the last 4 weeks, this blood will not need to be drawn. Women who are able to have children must have a negative blood (about 1 teaspoon) blood test within 2 weeks of study entry.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 3 groups.

If you are assigned to Group 1, you will receive TIV alone. If you are assigned to Group 2, you will receive pegylated interferon with TIV. If you are assigned to Group 3, you will receive interferon with TIV.

You will have an equal chance of being assigned to any of the 3 groups. Your doctor, the study doctor, study staff, and you will know which group you are in.

Study Drug Administration:

You will receive TIV through a needle into a muscle in your arm (the arm you do not write with) on Days 1 and 28.

* If you are in Group 1, you will only receive TIV
* If you are in Group 2, you will receive pegylated interferon right before you receive TIV. It will be given through a needle under the skin. It will be given near the TIV injection site.
* If you are in Group 3, you will receive interferon right before you receive TIV. It will be given through a needle under the skin. It will be given near the TIV injection site.

After you are given the injection(s), you will be watched for 15 minutes in the clinic before you are allowed to go home.

You will keep a diary for 1 week (7 days) after the injection(s). In it, you will record any symptoms you may be experiencing, and you will also record your body temperature.

Study Visits:

On Day 1, blood (about 4 teaspoons) will be drawn to check your immune system's response to the flu virus.

On Day 8, you will be asked to return to the clinic and your symptom/temperature diary will be reviewed. If you cannot come to the clinic, a member of the research staff will call you to review this information. This phone call will take 15-30 minutes.

On Day 28, blood (about 4 teaspoons) will be drawn to check your immune system response to the flu virus.

On Day 56, blood (about 4 teaspoons) will be drawn to check you immune system response to the flu virus. If you live out of town and cannot return to M. D. Anderson for this visit, you may have your blood drawn at a local clinic. You will then mail the blood to the study doctor in a pre-paid envelope.

On Month 6, you will be called and asked about any side effects you may have experienced. This phone call will take 15-30 minutes.

Length of Study:

You will be considered off study after the Month 6 phone call. You will be taken off-study early if intolerable side effects or an allergic reaction occurs.

This is an investigational study. TIV, pegylated interferon, and interferon are FDA approved and commercially available. At this time, the use of pegylated interferon and standard interferon with TIV is only being used for research.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the protocol requirements and risks and providing written informed consent.
2. Patients with histologically or cytologically confirmed diagnosis of chronic lymphocytic leukemia according to established guidelines.
3. Patients with Rai stages 0 to 4.
4. Age >/= 18 years old.
5. If patients have been treated with antineoplastic therapy, it must have been finished 3 months or longer prior to enrollment.
6. Patients with complete or partial remission and those with stable (CLL) disease will be considered.
7. Patients who have received influenza vaccine in past 4 months will also be considered.
8. Patients willing to receive recombinant cytokine.
9. Patient willing to receive commercially available influenza vaccine that will not provide protection against the following years of influenza strains.
10. Patients must have adequate hepatic function defined as follows: total bilirubin </= 2.0 mg/dL; SGOT and /or SGPT </= 3 x upper normal limit of the reference laboratory value unless liver function abnormalities are considered due to underlying cancer or congenital hemolytic disorders.
11. Patient should avoid H2 blockers while on study. However, if H2 blockers are required to use, this will be reported and will be taken in consideration during response rate analysis.
12. Females patients who are able to have children must agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control during the time period starting 2 weeks prior to enrollment through 1 month from last vaccination dose. Acceptable methods of birth control are: intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge and condom. If they suspect pregnancy during the study, they must notify the study doctor.

Exclusion Criteria:

1. Concurrent serious medical illness in the opinion of Principle Investigator that could potentially interfere with protocol compliance.
2. Concurrent or previous malignancy whose prognosis is poor (< 90% probability of survival is 5 years).
3. History of known chronic viral infections within 12 months, including HIV and Hepatitis B or Hepatitis C. A screening for hepatitis or HIV will not be performed for this study.
4. Positive screening pregnancy test within 2 weeks in non-menopausal women or breast-feeding.
5. Patients with known allergy to either vaccine or interferon preparation.
6. Patients with neutropenia (ANC < 500 cells/uL) within 4 weeks.
7. Patients with lymphocytopenia (ALC < 300 cells/uL) within 4 weeks.
8. Concomitant use of investigational vaccines and/or medications within four weeks prior to study entry, or expected use of experimental or licensed vaccines or blood/blood products prior to study completion.
9. Receipt of immunoglobulin in 3 months.
10. Subject is enrolled in a conflicting clinical trial.
11. History of Guillain-Barre Syndrome.
12. Has an acute illness including an oral temperature greater than 100.4°F, within one week of vaccination.
13. In patients who have prior therapy with fludarabine or alemtuzumab (Campath®), the treatment must have completed 12 months prior to enrollment.
14. In patients who have prior therapy with Rituximab (Rituxan®), the treatment must have completed 6 months prior to enrollment.
15. Patients with history of medically significant psychiatric disease, especially endogenous depression (not reactive to diagnosis of cancer), psychosis and bipolar disorder.
16. Patients with seizure disorders requiring anticonvulsant therapy.
17. Patients with history of severe cardiac disease with New York Heart Association (NYHA) grade 3 or 4.
18. Patients with severe renal disease requiring hemodialysis.
19. Patients who have received H2 blockers such as Ranitidine, Cimetidine, or Famotidine within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04

PRIMARY OUTCOMES:
Immunogenicity rate | Day 1, 8, 28, 56 and 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Amar Safdar, MD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org